CLINICAL TRIAL: NCT02424344
Title: A Multiple Dose, Randomized, Double-blind, Placebo Controlled, Parallel Clinical Trial to Assess the Effect of Aclidinium Bromide/Formoterol Fumarate Fixed-dose Combination on Lung Hyperinflation, Exercise Capacity and Physical Activity in Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of Aclidinium/Formoterol on Lung Hyperinflation, Exercise Capacity and Physical Activity in Moderate to Severe COPD Patients
Acronym: ACTIVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6570C00001; M-40464-33 (Other: Clinical Trial Protocol Code); 2014-005318-50 (EudraCT Number)
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclidinium Bromide/Formoterol Fumarate FDC 400/12μg (Experimental): 8 weeks, double blind treatment period
  Interventions: Drug: Aclidinium/Formoterol
- Placebo to Aclidinium/Formoterol (Placebo Comparator): 8 weeks, double blind treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium/Formoterol — Aclidinium bromide/Formoterol fumarate FDC 400/12μg dry powder for oral inhalation twice daily via Genuair inhaler
  Arms: Aclidinium Bromide/Formoterol Fumarate FDC 400/12μg
Drug: Placebo — Dose-matched placebo dry powder for oral inhalation twice daily via Genuair inhaler
  Arms: Placebo to Aclidinium/Formoterol

SUMMARY:
The present study is planned to evaluate the effect of the aclidinium bromide/formoterol fumarate 400/12 μg FDC BID on the hyperinflation, exercise endurance and physical activity in patients with moderate to severe COPD. Additionally, the effect of the behavioural intervention on top of aclidinium bromide/formoterol fumarate 400/12 μg will be assessed both on the exercise endurance and the physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant, non-lactating females aged ≥ 40.
2. Patients with a clinical diagnosis of COPD according to GOLD guidelines 2014, with a post bronchodilator FEV1 ≥ 40% and < 80% of the predicted value and FEV1/FVC < 70% at Visit 1.
3. Functional residual capacity (FRC) measured by body plethysmography at Visit 1 ≥ 120% of predicted value.
4. Patients with modified Medical Research Council dyspnea scale (mMRC) ≥ 2 at Visit 1.
5. Current or former cigarette smokers with a smoking history of at least 10 pack-years at Visit 1
6. Patients willing to participate in the telecoaching program during the four last weeks and to enhance their physical activity
7. Patients who understand and are able to follow the study procedures, are cooperative and are willing to participate in the study as indicated by signing the informed consent.

Exclusion Criteria:

1. History or current diagnosis of asthma.
2. Any respiratory tract infection (including upper respiratory tract) or COPD exacerbation in the 6 weeks prior to Visit 1 or during the run-in period.
3. Patients who have been hospitalised for an acute COPD exacerbation within 3 months prior to Visit 1 or during the run-in period.
4. Clinically significant respiratory conditions other than COPD.
5. Use of long-term oxygen therapy (≥ 15 hours/day).
6. Oxygen saturation ≤ 85% as measured by pulse oximetry during exercise testing at Visit 1, Visit 2 or Visit 3 prior to randomisation.
7. Patients with a Body Mass Index (BMI) ≥ 40kg/m2.
8. Patient who may need to start a pulmonary rehabilitation program during the study and/or who started/finished it within 3 months prior to Visit 1 or during the run-in period.
9. Patients with clinically significant cardiovascular conditions.
10. Patients with Type I or uncontrolled Type II diabetes, uncontrolled hypo-or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled or untreated hypertension.
11. Patient with known non-controlled history of infection with human immunodeficiency virus (HIV) and/or active hepatitis.
12. Patients with clinically relevant abnormalities in the results of the blood pressure, ECG, or physical examination at Visit 1.
13. Patients with any serious or uncontrolled physical or mental dysfunction that could place the patient at higher risk derived from his/her participation in the study or could confound the results
14. Patients with conditions other than COPD that may contribute to dyspnoea and exercise limitation or with contraindications to clinical exercise testing according to ATS recommendations for CPET
15. Patients with other relevant comorbidities that make the patient nor suitable to follow-up study procedures and/or could affect physical activity
16. Patients who cycled < 2 minutes or > 15 minutes during the constant work-rate exercise tests conducted at Visit 2 (Run-in Visit) or at Visit 3 even after adjustment of the work load.
17. Patients with history of hypersensitivity reaction to inhaled anticholinergics, sympathomimetic amines or inhaled medication or any component thereof (including report of paradoxical bronchospasm)
18. Patients for whom the use of anticholinergic drugs is contraindicated (acute urinary retention, symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma)
19. Patients unable to properly use a multidose dry powder inhaler or a pressurized metered-dose inhaler (pMDI).
20. Patients using any prohibited medication (including IMP within 30 days (or 6 half-lives, whichever is longer) before Visit 1) or who have not undergone the required washout period.
21. History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer).
22. Patients who do not maintain regular day/night, waking/sleeping cycles (e.g., night shift workers, sleep apnea).
23. Patients unable to give their consent, or patients of consenting age but under guardianship, or vulnerable patients

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2016-07-25 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Canada (4):
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Sainte-Foy, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Germany (10):
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Jena
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Wiesbaden
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Nyíregyháza
  - Research Site, Törökbálint
- Spain (3):
  - Research Site, Alicante
  - Research Site, Cáceres
  - Research Site, Madrid

REFERENCES:
- [Derived] Koopman M, Franssen FME, Gaffron S, Watz H, Troosters T, Garcia-Aymerich J, Paggiaro P, Molins E, Moya M, van Burk L, Maier D, Garcia Gil E, Wouters EFM, Vanfleteren LEGW, Spruit MA. Differential Outcomes Following 4 Weeks of Aclidinium/Formoterol in Patients with COPD: A Reanalysis of the ACTIVATE Study. Int J Chron Obstruct Pulmon Dis. 2022 Mar 8;17:517-533. doi: 10.2147/COPD.S308600. eCollection 2022. PMID 35342289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 study centers, 15 in Germany, 4 in Hungary, 3 in Spain and 4 in Canada. The first patient was enrolled in April 2015 and the last patient visit was in July 2016.
Pre-assignment Details: 335 patients were screened; 267 were assessed as eligible and were randomized into the study. 68 patients failed screening. The main reason for screening failure was non-fulfilment of inclusion or exclusion criteria (16.7%).
Groups:
- AB/FF 400/12 μg: Aclidinium Bromide/Formoterol Fumarate 400/12 μg
- Placebo: Placebo to Aclidinium/Formoterol
Period: Overall Study
Arm/Group | AB/FF 400/12 μg | Placebo
Started | 134 | 133
Completed | 127 | 123
Not Completed | 7 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 4 | 8

BASELINE CHARACTERISTICS:
Population: The Safety Population defined as all randomized patients who took at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | AB/FF 400/12 μg | Placebo | Total
Number analyzed (Participants) | 134 | 133 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (7.9) | 62.1 (7.7) | 62.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 107
  Male | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Functional Residual Capacity (FRC) After 4 Weeks of Treatment
Description: Baseline values in FRC were defined as the corresponding values just before randomization on Day 1 of treatment (Week 0). Trough values were obtained prior to study drug administration.
Time Frame: Baseline and Week 4
Population: The intent-to-treat (ITT) population - equal to the Safety population and defined as all randomised patients who took at least one dose of investigational product (IP) - who had available trough FRC values at baseline and Week 4.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | AB/FF 400/12 μg | Placebo
Number analyzed (Participants) | 124 | 125
Liters | -0.162 (0.050) | -0.037 (0.050)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs Placebo; Test type: Superiority or Other; p = 0.069, ANCOVA; Adjusted by baseline and age as covariates, and treatment group, sex and smoking-status as fixed effect factors; Least Square mean difference = -0.125, 95% CI 2-sided [-0.259 to 0.010]

2. Secondary Outcome: Change From Baseline in Endurance Time (ET) During Constant Work Rate Cycle Ergometry at Week 8
Description: The ET was the time from the increase in work rate to 75% Wmax to the point of symptom limitation.
  Baseline measurements were taken prior to the IP dose on Day 1. Measurements at Week 8 were taken at 3 hours post-dose. Participants underwent a behavioural intervention (consisting of a telecoaching programme to enhance physical activity) between Week 4 and Week 8.
Time Frame: Baseline to Week 8
Population: Intention-to-treat population - which was equal to the safety population, defined as all participants who took at least one dose of investigational product - who had available ET values at baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | AB/FF 400/12 μg | Placebo
Number analyzed (Participants) | 124 | 121
Seconds | 50.7 (18.1) | -4.6 (18.2)

3. Secondary Outcome: Percentage of Inactive Patients (Mean of <6000 Steps Per Day) at Week 8
Description: Physical activity was assessed by means of measurement of activity parameters (e.g. number of steps) through a Dynaport MoveMonitor and completion of the Daily ProActive Physical Activity in chronic obstructive pulmonary disease (COPD) questionnaire.
  Compliant criterion based on at least 8 hours per day, and at least 3 days per week. Participants underwent a behavioural intervention (consisting of a telecoaching programme to enhance physical activity) between Week 4 and Week 8.
  Baseline was defined as mean of steps/day assessed during the week before the randomisation visit.
Time Frame: Week 8
Population: The intent-to-treat (ITT) population - equal to the Safety population and defined as all randomised patients who took at least one dose of IP
  - who had available activity data (compliant criterion).
Measure: Number; unit: Percent of inactive participants
Arm/Group | AB/FF 400/12 μg | Placebo
Number analyzed (Participants) | 118 | 117
Percent of inactive participants | 41.53 | 50.43

ADVERSE EVENTS:
Time Frame: From Screening, Week -2 (Days -17 to -11) to Follow-up, Week 10 (Day 70+3)
Arm/Group | AB/FF 400/12 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/134 | 3/133
Other Adverse Events (participants affected / at risk) | 14/134 | 24/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=134) | Placebo (N=133)
Fatigue (General disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=134) | Placebo (N=133)
Nasopharyngitis (Infections and infestations) | 14 (14) | 13 (13)
Headache (Nervous system disorders) | 4 (4) | 12 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Principal Investigator (PI) will be subject to mutual agreement between the PI and the sponsor.